CLINICAL TRIAL: NCT05217654
Title: A Randomized, Double - Blind, Placebo - Controlled Trial to Investigate the Effect of Dapagliflozin on Ischemia Reperfusion Induced Endothelial Dysfunction of the Forearm Vasculature in Healthy Male Subjects
Brief Title: Trial to Investigate the Effect of Dapagliflozin on Ischemia Reperfusion Induced Endothelial Dysfunction
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Wolzt, Prof. MD, Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: FBF-SGLT2
Record Dates: First submitted 2022-01-05; First posted 2022-02-01 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Reperfusion Injury; Vascular Complications
Keywords: dapagliflozin; forearm blood flow measurement; reperfusion injury; vascular function
MeSH Terms: conditions — Reperfusion Injury | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled, double-blind, parallel group, phase 1 trial. Subjects in study group A will receive a daily oral dose of 10 mg dapagliflozin for 14 days (until study day 15) Subjects in study group B will receive a 14 day treatment with placebo-dapagliflozin.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin (Active Comparator): 14 day orally treatment with dapagliflozin
  Interventions: Drug: Dapagliflozin 10mg
- Dapagliflozin-placebo (Placebo Comparator): 14 day orally treatment with dapagliflozin - placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Daily orally administration of 10mg dapagliflozin
  Other Names: Forxiga 10mg Tabletten
  Arms: Dapagliflozin
Drug: Placebo — Daily orally administration of 10mg dapagliflozin-placebo
  Other Names: Placebo tablets
  Arms: Dapagliflozin-placebo

SUMMARY:
The aim of the study is to investigate the effect of dapagliflozin or placebo on acetylcholine (Ach)- or nitroglycerin (GTN)-induced vasodilation of the forearm resistance vasculature, as determined by FBF measurement before and 10 minutes after 20 minutes of forearm ischemia.

DETAILED DESCRIPTION:
The aim is to test the effect of dapagliflozin or placebo on ACh-induced vasodilatation of the forearm resistance vasculature as assessed by FBF measurement before and 10 min after a 20 min forearm ischemia as well as after a 14 day treatment period. The area under the dose-effect curve (AUC) of different ACh doses will be calculated and compared between treatment groups (dapagliflozin vs. placebo) and different time points (pre-ischemia vs. post-ischemia). FBF measurements will be made in response to increasing intra-arterial doses of ACh (25, 50, 100 nmol/min) to assess endothelial function or GTN (4, 8, 16 nmol/min) to test vascular smooth muscle vasodilator function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects; 18 - 40 years of age
* Body mass index between 18 and 27 kg/m2
* Written informed consent
* Normal findings in medical history
* Non-smoking

Exclusion Criteria:

* Regular intake of any medication including OTC drugs and herbals within 2 weeks before IMP administration
* History of occlusive vascular diseases
* History of vascular anomalies
* History of coagulation disorders
* History of diabetes mellitus (Type 1&2) or pre-diabetes (i.e. HbA1c ≥ 5,7 %)
* History of kidney disease
* History of ketoacidosis
* Impaired liver function (AST, ALT, gGT, bilirubin >3 x ULN)
* Impaired renal function (serum creatinine > 1.3 mg/dl)
* Any other relevant deviation from the normal range in clinical chemistry, haematology or urine analysis
* HIV-1/2-Ab, HbsAg or HCV-Ab positive serology
* Systolic blood pressure above 145 mmHg, diastolic blood pressure above 95 mmHg
* Known allergy against any test agent under study and/or lactose intolerance
* Regular daily consumption of more than on litre of xanthine-containing beverages or more than 40g alcohol
* Participation in another clinical trial during the preceding 3 weeks

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-02-18 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Acetylcholine - Area under the curve forearm blood flow measurement | 14 days
  effect of dapagliflozin after a two weeks period of regular intake on forearm blood flow (FBF) reactivity in response to the vasodilators acetylcholine (ACh; endothelium-dependent agonist) or nitroglycerin (GTN; endothelium-independent vasodilator)
Acetylcholine - Area under the curve forearm blood flow measurement | 30 min
  acute effect of dapagliflozin on forearm blood flow (FBF) reactivity in response to the vasodilators acetylcholine (ACh; endothelium-dependent agonist) or nitroglycerin (GTN; endothelium-independent vasodilator) 10 min before (baseline) and after 20 min forearm ischemia, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eltzschig HK, Eckle T. Ischemia and reperfusion--from mechanism to translation. Nat Med. 2011 Nov 7;17(11):1391-401. doi: 10.1038/nm.2507. PMID 22064429
- [Background] Szabo C. The pathophysiological role of peroxynitrite in shock, inflammation, and ischemia-reperfusion injury. Shock. 1996 Aug;6(2):79-88. doi: 10.1097/00024382-199608000-00001. PMID 8856840
- [Background] Pleiner J, Schaller G, Mittermayer F, Marsik C, MacAllister RJ, Kapiotis S, Ziegler S, Ferlitsch A, Wolzt M. Intra-arterial vitamin C prevents endothelial dysfunction caused by ischemia-reperfusion. Atherosclerosis. 2008 Mar;197(1):383-91. doi: 10.1016/j.atherosclerosis.2007.06.011. Epub 2007 Jul 23. PMID 17645881
- [Background] Lu Q, Liu J, Li X, Sun X, Zhang J, Ren D, Tong N, Li J. Empagliflozin attenuates ischemia and reperfusion injury through LKB1/AMPK signaling pathway. Mol Cell Endocrinol. 2020 Feb 5;501:110642. doi: 10.1016/j.mce.2019.110642. Epub 2019 Nov 21. PMID 31759100
- [Background] Korkmaz-Icoz S, Kocer C, Sayour AA, Kraft P, Benker MI, Abulizi S, Georgevici AI, Brlecic P, Radovits T, Loganathan S, Karck M, Szabo G. The Sodium-Glucose Cotransporter-2 Inhibitor Canagliflozin Alleviates Endothelial Dysfunction Following In Vitro Vascular Ischemia/Reperfusion Injury in Rats. Int J Mol Sci. 2021 Jul 21;22(15):7774. doi: 10.3390/ijms22157774. PMID 34360539
- [Background] Khemais-Benkhiat S, Belcastro E, Idris-Khodja N, Park SH, Amoura L, Abbas M, Auger C, Kessler L, Mayoux E, Toti F, Schini-Kerth VB. Angiotensin II-induced redox-sensitive SGLT1 and 2 expression promotes high glucose-induced endothelial cell senescence. J Cell Mol Med. 2020 Feb;24(3):2109-2122. doi: 10.1111/jcmm.14233. Epub 2019 Mar 30. PMID 30929316
- [Background] Tsai KL, Hsieh PL, Chou WC, Cheng HC, Huang YT, Chan SH. Dapagliflozin attenuates hypoxia/reoxygenation-caused cardiac dysfunction and oxidative damage through modulation of AMPK. Cell Biosci. 2021 Feb 26;11(1):44. doi: 10.1186/s13578-021-00547-y. PMID 33637129
- [Background] He C, Zhu H, Li H, Zou MH, Xie Z. Dissociation of Bcl-2-Beclin1 complex by activated AMPK enhances cardiac autophagy and protects against cardiomyocyte apoptosis in diabetes. Diabetes. 2013 Apr;62(4):1270-81. doi: 10.2337/db12-0533. Epub 2012 Dec 7. PMID 23223177
- [Background] Chen X, Li X, Zhang W, He J, Xu B, Lei B, Wang Z, Cates C, Rousselle T, Li J. Activation of AMPK inhibits inflammatory response during hypoxia and reoxygenation through modulating JNK-mediated NF-kappaB pathway. Metabolism. 2018 Jun;83:256-270. doi: 10.1016/j.metabol.2018.03.004. Epub 2018 Mar 9. PMID 29526538
- [Background] Liem DA, Verdouw PD, Duncker DJ. Transient limb ischemia induces remote ischemic preconditioning in vivo. Circulation. 2003 Jun 24;107(24):e218-9; author reply e218-9. doi: 10.1161/01.CIR.0000077520.36997.F9. No abstract available. PMID 12821595
- [Background] Kharbanda RK, Peters M, Walton B, Kattenhorn M, Mullen M, Klein N, Vallance P, Deanfield J, MacAllister R. Ischemic preconditioning prevents endothelial injury and systemic neutrophil activation during ischemia-reperfusion in humans in vivo. Circulation. 2001 Mar 27;103(12):1624-30. doi: 10.1161/01.cir.103.12.1624. PMID 11273988
- [Background] Benjamin N, Calver A, Collier J, Robinson B, Vallance P, Webb D. Measuring forearm blood flow and interpreting the responses to drugs and mediators. Hypertension. 1995 May;25(5):918-23. doi: 10.1161/01.hyp.25.5.918. PMID 7737727
- [Background] Barcroft H, Edholm OG. The effect of temperature on blood flow and deep temperature in the human forearm. J Physiol. 1943 Jun 30;102(1):5-20. doi: 10.1113/jphysiol.1943.sp004009. No abstract available. PMID 16991588
- [Background] Seman L, Macha S, Nehmiz G, Simons G, Ren B, Pinnetti S, Woerle HJ, Dugi K. Empagliflozin (BI 10773), a Potent and Selective SGLT2 Inhibitor, Induces Dose-Dependent Glucosuria in Healthy Subjects. Clin Pharmacol Drug Dev. 2013 Apr;2(2):152-61. doi: 10.1002/cpdd.16. Epub 2013 Mar 27. PMID 27121669
- [Background] Fralick M, Schneeweiss S, Patorno E. Risk of Diabetic Ketoacidosis after Initiation of an SGLT2 Inhibitor. N Engl J Med. 2017 Jun 8;376(23):2300-2302. doi: 10.1056/NEJMc1701990. No abstract available. PMID 28591538
- [Background] Weisshaar S, Litschauer B, Kerbel T, Wolzt M. Atorvastatin combined with ticagrelor prevent ischemia-reperfusion induced vascular endothelial dysfunction in healthy young males - A randomized, placebo-controlled, double-blinded study. Int J Cardiol. 2018 Mar 15;255:1-7. doi: 10.1016/j.ijcard.2017.12.067. Epub 2017 Dec 24. PMID 29288055
- [Background] Weisshaar S, Litschauer B, Eipeldauer M, Hobl EL, Wolzt M. Ticagrelor mitigates ischaemia-reperfusion induced vascular endothelial dysfunction in healthy young males - a randomized, single-blinded study. Br J Clin Pharmacol. 2017 Dec;83(12):2651-2660. doi: 10.1111/bcp.13378. Epub 2017 Aug 22. PMID 28715608
- [Derived] Lutnik M, Weisshaar S, Litschauer B, Bayerle-Eder M, Niederdockl J, Wolzt M. Dapagliflozin prevents vascular ischemia-reperfusion injury in healthy young males: a randomized, placebo-controlled, double-blinded trial. Sci Rep. 2025 May 13;15(1):16633. doi: 10.1038/s41598-025-01405-4. PMID 40360700